CLINICAL TRIAL: NCT04658706
Title: Supervised Exercise for Head and Neck Cancer Patients Initiated Previously or After Treatment: the SEHNeCa Randomized Controlled Trial
Brief Title: The SEHNeCa Supervised Exercise Project
Acronym: SEHNeCa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Jon Cacicedo Fernandez Bobadilla, Principal investigator, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PI 20/00112
Record Dates: First submitted 2020-11-25; First posted 2020-12-08 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-02

CONDITIONS: Neack and Head Cancer; Supervised Execise Program
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Sham Comparator): a physical activity prescription to be performed autonomously
  Interventions: Other: exercise prescription
- Prehabilitation (Experimental): They will receive a supervised exercise programat least 2 weeks before starting the conventional chemoradiotherapy treatment and concomitant
  Interventions: Other: A supervised exercise program
- Rehabilitation (Experimental): They will receive a supervised exercise programat 12 weeks after the first radiotherapy session, once standard treatment has finished
  Interventions: Other: A supervised exercise program

INTERVENTIONS:
Other: A supervised exercise program — is a 12-week exercise program supervised by specially trained instructors combining moderate to high intensity aerobic and strength exercises (three 1 hour sessions a week).
  Arms: Prehabilitation; Rehabilitation
Other: exercise prescription — they will receive a prescription concerning healthy lifestyles and a personalized exercise plan
  Arms: Control

SUMMARY:
Objectives:

* To evaluate the effectiveness and efficiency of an innovative supervised exercise program for patients with head and neck cancer (SEHNeCa) to ameliorate loss of lean body mass, functional capacity and quality of life during one year, compared to a reference group receiving a physical activity prescription to be performed autonomously.
* To identify the optimal timing for applying the supervised exercise program: in a Prehabilitation period, at least 2 weeks before starting the conventional chemoradiotherapy treatment and concomitant with it, or during a Rehabilitation period, starting 12 weeks after the first radiotherapy session, once standard treatment has finished. Design: a multicenter, randomized clinical trial, where patients will be randomized to 3 groups: one control group and 2 experimental with different timing of exercise intervention. Population: 120 patients diagnosed with histological locally advanced stage III-IVa-b with squamous cell carcinomas of the larynx, pharynx, oral cavity, salivary or in neck lymph nodes from an unknown primary tumour treated with curative intent undergoing radiotherapy with or without concomitant chemotherapy.

SEHNeCa program: is a 12-week exercise program supervised by specially trained instructors combining moderate to high intensity aerobic and strength exercises (three 1 hour sessions a week). Outcome measurements: main outcome variable: change in body mass index at 6 months (multy-frecuenciy imoediance). Secondary variables at basal, 7, 12, 25, and 52 weeks after the beginning of radiotherapy include quality of life (general SF-36 and cancer specific quality of life -European Organization for Research and Treatment of Cancer QLQ-C-30-),functional capacity (6 min walking test), patient reported outcomes and treatment maximum adverse events. Analyses: Differences between treatment groups in changes in outcome variables will be analyzed on an intention to treat basis. We will use linear mixed models for longitudinal analysis of repeated measurements of continuous outcomes (SAS PROC MIXED) and generalized logistic mixed models for dichotomous (SAAS PROC GLIMMIX), considering intercept and time courses as random effects and testing the significance of the interaction of time slopes by treatment group.

ELIGIBILITY:
Inclusion Criteria:

Histological diagnosed locally advanced stage III-IVa-b with squamous cell carcinomas of the larynx, pharynx, oral cavity, salivary or in neck lymph nodes from an unknown primary tumour (TNM 9th AJCC classification; 2019.) treated with curative intent undergoing radiotherapy with or without concomitant chemotherapy (with or without previous surgery).

* Age: more than 18 years
* WHO performance status of 0-1 (IK 80%)
* Body mass index: more than 18.5.
* No evidence of metastatic disease
* No excessive alcohol intake (men > 21 and women > 14 units/week)
* No current or previous malignancies that could prevent participation and training
* No recent systematic resistance training.

Exclusion Criteria:

* Decompensated heart disease, uncontrolled hypertension (TAS>200 o TAD>110), cardiac insufficiency (NYHA II o mayor), heart failure or constrictive pericarditis, Neutropenia, severe anemia ( Hb<8.0 g/dl), platelets count <50.000 microL
* Other health problems in which exercise is contraindicated.
* Carry out physical activity regularly (150 min/week of moderate activity or 75 of vigorous activity), measured with the PVS questionarie.
* Pregnancy
* Tracheostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in body lean mass | Measured at baseline 7, 12, 25, and 52 weeks after the beginning of radiotherapy
  change in body lean mass will be measured at baseline 7, 12, 25, and 52 weeks after the beginning of radiotherapy) by the multi-frequency impedance measurement technique.

SECONDARY OUTCOMES:
Change in Quality of life | Measured at baseline 7, 12, 25, and 52 weeks after the beginning of radiotherapy
  evaluated with the EORTCQLQ-C-30 questionnaire associated with the head and neck 35 specific module. Cancer specific quality of life is evaluated by the European Organisation for Research and Treatment of Cancer (QLQ-C-30) questionnaire (Aaronson et al., 1993). The QLQ-C-30 questionnaire includes five functional domains (physical, role, cognitive, emotional and social; higher scores represent greater function/quality of life) and three symptom scales (fatigue, pain and nausea; lower scores represent greater quality of life/less symptom severity)
Change in Functional capacity | Measured at baseline 7, 12, 25, and 52 weeks after the beginning of radiotherapy
  Evaluated by the six minute walking test
Change in Strenght | Measured at baseline 7, 12, 25, and 52 weeks after the beginning of radiotherapy
  Evaluated by a manual dynamometer for higher body and by the bench press for the lower body
Change in Quality of life | Measured at baseline 7, 12, 25, and 52 weeks after the beginning of radiotherapy
  Evaluated by the Medical Outcomes Study 36- Item Short-Form Health Survey (SF-36). The HRQL questionnaire is measured blindly with self-administered questionnaires: the Spanish version of the SF-36 and. Questionnaire will be filled out before and after the intervention. SF-36 generates an 8-dimension health profile and two summary scores for the physical and mental components. This questionnaire has been validated in the Spanish population.
Change in Functional capacity | Measured at baseline 7, 12, 25, and 52 weeks after the beginning of radiotherapy
  Evaluated by the shoulder pain disability index. patients place a mark on a 10cm visual analogue scale for each question. Verbal anchors for the pain dimension are 'no pain at all' and 'worst pain imaginable', and those for the functional activities are 'no difficulty' and 'so difficult it required help'. The scores from both dimensions are averaged to derive a total score. As more score, more pain the patients feels.
Change in Functional capacity | Measured at baseline 7, 12, 25, and 52 weeks after the beginning of radiotherapy
  Evaluated by Fatigue-related measure with the FACIT-F test Predictor. a 13 items scale that measures the cancer related fatigue. The FACT-G scoring guide identifies those items that must be reversed before being added to obtain subscale totals. Negatively stated items are reversed by subtracting the response from "4". After reversing proper items, all subscale items are summed to a total, which is the subscale score.The higher score the score, the better the QOL.

CONTACTS AND LOCATIONS:
Locations (1):
- Biocruces Bizkaia research health institute, Barakaldo, Bizkaia, Spain

REFERENCES:
- [Derived] Rodriguez-Arietaleanizbeaskoa M, Mojas Ereno E, Arietaleanizbeaskoa MS, Grandes G, Rodriguez Sanchez A, Urquijo V, Hernando Alday I, Dublang M, Angulo-Garay G, Cacicedo J; SEHNeCa group. Protocol for the SEHNeCa randomised clinical trial assesing Supervised Exercise for Head and Neck Cancer patients. BMC Cancer. 2023 Mar 24;23(1):271. doi: 10.1186/s12885-023-10718-4. PMID 36964485